CLINICAL TRIAL: NCT00271349
Title: Budesonide for Eosinophilic Esophagitis: a Randomized, Placebo-controlled, Double-blind Treatment Study
Brief Title: Budesonide for Eosinophilic Esophagitis
Acronym: BEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss EE Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5257L00017; D5257L00017
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2009-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Budesonide
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide

SUMMARY:
Eosinophilic Esophagitis (EE) is a chronic, T-helper 2 cell (TH2) - type inflammatory disorder of the esophagus with a rapidly increasing prevalence. Studies analyzing the natural course of EE provide strong evidence, that the chronic inflammation leads to irreversible structural changes in the esophagus with a loss of the mucosal elasticity and a fibrosis of the sub-epithelial esophageal layers with a concomitant risk of impairment in function.

Treatment strategies in chronic inflammations have, in general, two main goals: 1) Relief of symptoms and 2) Prevention of long-term damage of the affected organ. Until now, the treatment of EE is still controversial. Standard recommendations for therapy of this chronic eosinophilic inflammation include dilation, systemic or topical corticosteroids and leukotriene antagonists. Several of these reports demonstrate, that topical corticosteroids may be effective for symptom control as well as for down-regulating the local inflammation. Furthermore it has been demonstrated, that treatment with topical corticosteroids is as effective as oral prednisone. However, the majority of therapeutic recommendations are based on clinical observations, case reports or small case series.

The purpose of this study is the evaluation of the efficacy and the safety of a monotherapy with a topical corticosteroid as short-term induction-treatment and as long-term, maintenance-treatment compared with placebo, in the treatment of adult patients with active EE.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, single center clinical trial to evaluate the efficacy and safety of topically applied Budesonide in the treatment of adult patients with Eosinophilic Esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Isolated Eosinophilic Esophagitis
* Adult patients (age > 14 years)
* Active disease (clinically and histologically)
* Informed Consent

Exclusion Criteria:

* Current use of specific treatments for EE
* Secondary causes of esophageal eosinophilia
* Intolerance to Budesonide
* Concomitant therapies for any reason that may affect assessment
* Use of an investigational drug with 30 days of entering the study
* Recent history or suspicion of current drug abuse and alcohol abuse
* Positive serum pregnancy test at the screening visit
* Any unstable serious co-existing medical condition

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-12; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of Budesonide in inducing a reduction of the esophageal eosinophilic infiltration in adult individuals with active EE after 2 weeks of induction-treatment.
Efficacy of Budesonide in sustaining a reduction of the esophageal eosinophilic infiltration in adult individuals with quiescent EE after 50 weeks of maintenance-treatment.

SECONDARY OUTCOMES:
Efficacy of Budesonide in inducing a reduction of the clinical manifestations of active EE after 2 weeks of induction-treatment.
Efficacy of Budesonide in sustaining a reduction of the clinical manifestations of quiescent EE after 50 weeks of maintenance-treatment.
Efficacy of a one year treatment with Budesonide on esophageal remodeling in adult subjects with EE.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Study Chair — Department of Gastroenterology, University Hospital Basel, Switzerland; Hans-Uwe Simon, MD, PhD, Study Director — Department of Pharmacology, University of Bern, Switzerland; Alex Straumann, MD, Principal Investigator — Department of Gastroenterology, Kantonsspital Olten, Switzerland
Locations (1):
- Department of Gastroenterology, Kantonsspital, Olten, Canton of Solothurn, Switzerland